CLINICAL TRIAL: NCT00237562
Title: Single Visit Cervical Cancer Prevention Program
Brief Title: Feasibility of the Management of Severe Cervical Dysplasia in a Single Visit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01CA076501 (NIH)
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2005-10

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

INTERVENTIONS:
Procedure: Large loop electrosurgical excision

SUMMARY:
1. Implement a single-visit program (SVP) for cervix cancer prevention in clinics serving a multi-ethnic population of women;
2. Set up an efficient system for interpretation of Pap smears for patients in the SVP that will minimize waiting time;
3. Determine the follow-up rates and compare them between women assigned to the SVP and a usual care program (UCP);
4. Determine satisfaction and compare it between women assigned to the SVP and the UCP;
5. Determine the cost-effectiveness and compare it between the SVP and UCP

DETAILED DESCRIPTION:
Women were recruited from underserved communities to participate in this single visit cervix cancer project. Large loop electrosurgical excision procedure (LEEP) was performed on SVP subjects with either a diagnosis of HGSIL/AGUS or suspicion of carcinoma. All other subjects with abnormal Papanicolaou smears were referred to our abnormal cytology clinics or received care in the community.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* No history of invasive cervical cancer
* Not pregnant

Exclusion Criteria:

* Absence of a cervix
* Abnormal vaginal bleeding
* Cervical cancer screening within the previous 12 months
* A known bleeding disorder
* Reluctance to be randomized
* Unwillingness to follow the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Manetta, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Orange, California, United States

REFERENCES:
- [Result] Brewster WR, Hubbell FA, Largent J, Ziogas A, Lin F, Howe S, Ganiats TG, Anton-Culver H, Manetta A. Feasibility of management of high-grade cervical lesions in a single visit: a randomized controlled trial. JAMA. 2005 Nov 2;294(17):2182-7. doi: 10.1001/jama.294.17.2182. PMID 16264159